CLINICAL TRIAL: NCT04859192
Title: Effect of Gamified Flipped Class Room on Facilitating Nursing Students' Skills Competency and Confidence
Brief Title: Gamified Flipped Class Room and Nursing Students' Skills Competency and Confidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, mohamed elsayed hamed elzeky, lecturer at medical surgical nursing faculty of nursing mansoura university, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MansouraN
Record Dates: First submitted 2021-04-19; First posted 2021-04-26 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Gamified Flipped Classroom; Education, Nursing Students

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): For 6 weeks, students in study group will receive their routine flipped classroom in addition to gamified activities that they are required to complete before class session.
  Interventions: Other: gamified flipped classroom
- control group (No Intervention): The control group will not receive any intervention only their routine flipped classroom education

INTERVENTIONS:
Other: gamified flipped classroom — moodle will be gamified
  Arms: study group

SUMMARY:
one of the primary components of effective teaching is student engagement and that engagement is critical for learning

DETAILED DESCRIPTION:
In order to increase motivation, it is necessary to eliminate the factors that create boredom and to transform the lectures into a more enjoyable environment. In recent years, the gamification strategy has been used in order to intrigue the students, and to increase their motivation for learning. Gamification is a system that implements game design components on out-of-game contexts and alters the subjects' behaviors.

ELIGIBILITY:
Inclusion Criteria:

* agree to participate.
* Registered fundamental II in second semester year (2020-2021).
* Have access to network at home.

Exclusion Criteria:

* • Previously enrolled in fundamental II course

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
changes in students learning motivation score | will be measured at baseline and at the end of study (after 6 weeks)
  will be measured using instructional material motivation survey.It consists of four domains: attention, relevance, confidence, and satisfaction, with a total of 36 questions on a 5-point Likert scale
change in skill practice confidence level | will be measured at baseline and at the end of study (after 6 weeks)
  confidence scale will be used to used to measure a student's confidence level related to skills performance
change in nursing students funadamental skill competency | will be measured at baseline and at the end of study (after 6 weeks)
  will be measured using observation checklist. it consists of eiight checklist and each checklist cover different nursing procedure. The evaluation items will be rated on a 3-point Likert scale
changes in students fundamental of nursing knowledge level | at baseline and three weeks and 6 weeks of study
  3 quizes,each composed of 20 questions. quiz 1 will measure students knowledge level at baseline on the first two procedures and quiz 2 and three will meassure knowledge level post implementation of gamified activitis after each three skills.

SECONDARY OUTCOMES:
intensity of nursing skills preparation | will be measured at baseline and at the end of study (after 6 weeks)
  three items which cover how often participants watched the skill video

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elzeky MEH, Elhabashy HMM, Ali WGM, Allam SME. Effect of gamified flipped classroom on improving nursing students' skills competency and learning motivation: a randomized controlled trial. BMC Nurs. 2022 Nov 16;21(1):316. doi: 10.1186/s12912-022-01096-6. PMID 36384544